CLINICAL TRIAL: NCT00155519
Title: A Psychopathological Study of Latent (Early) Schizophrenia: Clinical Pathology/Neuropsychological Dysfunctions
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 10892; NSC-89-2413-H-002-042; NSC-90-2413-H-0052-023
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-11-28 (Estimated); Status verified 2000-08

CONDITIONS: Schizophrenia; Latent Schizophrenia
Keywords: Schizophrenia; Latent Schizophrenia; Schizotypal Disorder; Psychopathology; Neuropsychological Function; Family History; Nosology; basic symptoms
MeSH Terms: conditions — Schizophrenia; Schizotypal Personality Disorder

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Current diagnostic criteria of schizophrenia are based on marked positive and negative symptoms. This definition may impede the exploration of basic phenomenological psychopathology or pathological mechanism of schizophrenia. Schizophrenia was found to have neuroanatomical, neurophysiological and neuropsychological impairment. However, the existence of these basic pathological states may not manifest as clinical state of schizophrenia, and it is found in normal relatives of schizophrenia proband. The clinical state of this underlying pathology may include so-called latent or early, or pseudo-neurotic schizophrenia or schizotypal disorder. The manifestation of prominent neurotic symptom state may not only present as an psychopathological issue, but also induce misdiagnosis in clinical practice. This may interfere early diagnosis of schizophrenia and may delay the chance of early and appropriate treatment.

Taking the fact of this disadvantaged conditions, this research is for exploration of clinical pathology and neuropsychological functions of latent or pseudo-neurotic schizophrenia. The strategy ia a natural follow-up study on the clinical cases obtained from the registration record of the medical charts of the National Taiwan University Hospital from 1970 to 1995. The natural follow-up results till study time (5 yrs to 30 yrs following period) will be explored. By using neurotic group (50 cases), latent schizophrenia group (50 cases) and schizotypal group (30 cases), the differences in clinical pathology, neuropsychological functions and family history of schizophrenia will be examined. There are 5 hypotheses to be tested: (1) Schizotaxia may exist as the manifestations of latent schizophrenia, schizotypal disorder and frank schizophrenia. The severity of pathology increased step by step; (2) The syndrome may change from the lower order to higher order to higher order, but not all of them changed to the higher order; (3) The clinical pathology of latent schizophrenia has both neurotic symptom as well as basic symptoms of schizophrenia; (4) There is the same kind of neuropsychological impairment of schizophrenia in the group of latent schizophrenia, and (5) The prevalence of schizophrenia in the first degree relatives of latent schizophrenia is higher than that of the general population. Finally, this study results will help the establishment of valid screening and/or diagnostic method (criteria) of latent schizophrenia for clinical and research usage.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia
* Latent Schizophrenia

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130
Dates: Start 2002-07; Study Completion 2002-07

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Gwo Hwu, Professor, Principal Investigator — National Taiwan University